

## CONSENT FORM FOR THE PARTICIPANT AND THE REPRESENTATIVE

Project title: MOVIE- Understanding viral load clearance in Mpox-positive patients.

Name of Principal Investigator/Project Investigator:

Oriol Mitjà (FIF) and Hypolite Muhindo (UNIKIN)

Version 2.0 14/07/2025

| Declaration | | Please initial or print<br>your thumb* on each<br>box |
|---|---|---|
| I confirm that I have read and understood the dated information sheet (version) for the study mentioned above. I have had the opportunity to review the information, ask questions and get satisfactory answers. | | |
| I understand that my consent is voluntary and that time without giving any reason and without affecti | • | |
| I understand that the relevant sections of my/part during the study may be accessed by authorized in relevant to my participation in this research. I give to these records. | idividuals from UNIKIN and FIF, when | |
| I understand that data about me/from the particip repository or by sharing it directly with other rese from this information | | |
| I understand that the tissue sample collected from<br>swab samples) will be used to support further rese<br>anonymously with other researchers, for their ethi | earch in the future, and may be shared | |
| I authorize that a copy of this consent form, which<br>the participant, be made available to the Study Coc<br>only. | • • | |
| I agree that I/the participant should take part in the above-mentioned study. | | |
| Participant's or Representative's printed name | Signature of Participant/Representative Date (or fingerprint/mark if you can't sign) | |
| Printed name of the person obtaining consent | Signature of the person obtaining consent | Date |
| The participant/representative is not able to sign. provided and that the participant/representative h read or write) | | |
| Printed name of impartial witness* | Signature of an impartial witness* | Date |



Project title: TRACE - Assessing the transmission dynamics of MPXV in monkeypox cases and contacts and determining the secondary attack rate (SAR) in contacts of positive cases.

Name of Principal Investigator/Project Investigator:

Oriol Mitjà (FIF) and Hypolite Muhindo (UNIKIN)

Version 2.0 14/07/2025

| Declaration | | Please initial or print |
|---|---|---|
| Deciaration | | your thumb* on each |
| | | box |
| I confirm that I have read and understood the dated information sheet (version) for the study mentioned above. I have had the opportunity to review the information, ask questions and get satisfactory answers. | | |
| I understand that my consent is voluntary and that time without giving any reason and without affecti | | |
| I understand that the relevant sections of my particle collected during the study may be accessed by auth UNIKIN and FIF, when relevant to my participation people to have access to these records. | | |
| I understand that data about me/from the participant may be shared through a public data repository or by sharing it directly with other researchers, and that I will not be identifiable from this information | | |
| I understand that the tissue sample collected from me/the participant (including blood and swab samples) will be used to support further research in the future, and may be shared anonymously with other researchers, for their ethically approved projects | | |
| I authorize that a copy of this consent form, which the participant, be made available to the Study Coo only. | | |
| I agree that I/the participant should take part in the above-mentioned study. | | |
| Participant's or Representative's printed name | Signature of Participant/Representative Date (or fingerprint/mark if you can't sign) | |
| Printed name of the person obtaining consent | Signature of the person obtaining consent | Date |
| The participant/representative is not able to sign. As a witness, I confirm that all information about the trial has been provided and that the participant/representative has consented to participate (*required only if the participant/representative cannot read or write) | | |
| Printed name of impartial witness* | Signature of an impartial witness* | |

Participant ID Number: